CLINICAL TRIAL: NCT07209553
Title: "Smart Breaks" During Working Hours: Feasibility of an AI-Based Application to Enhance Well-Being Through Active Micro-Breaks Among Office Workers
Brief Title: AI-Powered Micro-Breaks at Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West University of Timisoara (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SmartBreaks
Record Dates: First submitted 2025-09-09; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Musculoskeletal Discomfort; Work-related Vigor
Keywords: feasibility study; occupational health; AI coach; microbreaks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention involved using the Mobi AI coach to set up and engage in active micro-breaks over five consecutive working days.
  Interventions: Device: Mobi

INTERVENTIONS:
Device: Mobi — Mobi is a conversational AI coach that serves as an occupational health coach for employees. Through coaching conversations, Mobi gets to know each employee and help them set micro-goals to work towards their overall health goal/objective. Mobi suggests small, personalized activities for the micro-breaks that align with these goals. To ensure ease of use it is integrated into Slack and MS Teams.

SUMMARY:
This study evaluates the feasibility of an online intervention based on artificial intelligence-the Movebite app integrated into the Slack platform-aimed at promoting engagement in micro-breaks involving physical activity, with the goal of enhancing workplace well-being and reducing musculoskeletal discomfort among remote workers.

DETAILED DESCRIPTION:
Remote and hybrid work have intensified sedentary behavior, increasing the risk of professional burnout and negatively affecting employee health. This study investigates the feasibility and accessibility of the Movebite app, an AI-based tool integrated into Slack, designed to encourage active micro-breaks. Through a one-arm, pre-test post-test design, we evaluate the feasibility and usability of the AI-based virtual coach and its relevance for well-being of employees working from home.

This research contributes to the development and promotion of empirically grounded solutions in the field of occupational health psychology, testing an innovative technological approach to reduce the negative impact of sedentary work.

ELIGIBILITY:
Inclusion Criteria:

* Employees between the ages of 18-60 years' old
* Full-time working entirely from home (home office)
* Have a PC or laptop and basic digital competencies
* Proficient in English language

Exclusion Criteria:

* Other work arrangements such as shift-work, part-time work
* Unable to access the internet/computer/install Slack app (Yes/No questions)
* No proficiency for English
* Not working mainly from a desk (e.g., fieldwork)
* Current health issues (current pregnancy, any neurological, vascular, or acute musculoskeletal condition or any disease or symptom)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the intervention | Post-intervention (1 week).
  Seven additional items are open-ended and will be analyzed qualitatively. These items allow participants to elaborate on what aspects of the program they found most or least valuable, describe their experience with communication tools within the intervention, and offer suggestions for improvement.
System usability | Post-intervention (1 week)
  We will use a 10 item questionnaire (Bangor et al., 2009) designed to measure participants' satisfaction with Mobi, the AI health coach. The total score of System Usability Scale is 0 and the highest one is 100. A higher score means a better outcome.
Treatment adherence | Post-intervention only (1 week)
  Dropout rate and frequency of app usage.
Vigor | Change from baseline to post-test (1 week; 5 workdays)
  Vigor refers to a positive affective state experienced at work. It will be assessed using five items from the Physical Strength subscale of the instrument developed by Shirom (2003). A higher score means a better outcome (i.e., increased employee vigor).
Focus | Change from baseline to post-test (1 week; 5 workdays).
  Focus refers to an employee's capacity to maintain attention and mental clarity while working. It will be assessed using five items from the Cognitive Liveliness subscale of the instrument developed by Shirom (2003). A higher score indicates a better outcome (i.e., increased cognitive focus at work).
Physical (dis)comfort | Change from baseline to post-test (1 week; 5 workdays)
  Physical discomfort (musculoskeletal pain) will be measured using a single-item instrument based on the Visual Analog Scale (VAS) (Häfeli & Elfering, 2006). The VAS is a widely used and validated method for assessing subjective physical symptoms such as pain intensity. Participants will indicate their level of discomfort by marking a point along a continuum, reflecting their experience over the past week. Higher scores indicate greater musculoskeletal discomfort.
Positive and negative affect | Change from baseline to post-test (1 week; 5 workdays)
  Affect will be measured using the Positive Affect subscale from the Positive and Negative Affect Schedule (PANAS; Watson, Clark, & Tellegen, 1988). This scale assesses the extent to which individuals have experienced a range of positive emotions (e.g., enthusiastic, inspired, alert) over the past week. Participants rate each item on a 5-point scale, from "Very slightly or not at all" to "Extremely." Higher scores reflect a higher level of positive emotional experience.

OTHER OUTCOMES:
Physical activity during work | Baseline only
  What employees currently do to stay active during working hours (i.e., stretching, short walks, taking the stairs, using a standing desk, scheduled workout sessions during work, other)
Before and/or after-work physical activities | Baseline only
  To assess participants' engagement in physical activity outside working hours, we included two binary (Yes/No) items referring to typical weekly behaviors. The first item evaluates whether participants engage in light movement after work hours (e.g., walking, stretching), while the second item assesses participation in regular, scheduled workout sessions either before or after the workday. These items aim to provide a brief overview of participants' physical activity routines that may contribute to their overall well-being and complement the effects of the intervention.
Sociodemographic information | Baseline only
  Age, gender, background, educational level, average monthly income, work experience, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- West University of Timisoara, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bangor, A., Miller, J. & Kortum, P. (2009). Determining what individual SUS scores mean: Adding an adjective rating scale. Journal of Usability Studies, 4(3), 114-123. Retrieved from http://uxpajournal.org/determining-what-individual-sus-scores-mean-adding-an-adjective-rating-scale/
- [Background] Shirom, A. (2003). Feeling vigorous at work? The construct of vigor and the study of positive affect in organizations. In Emotional and physiological processes and positive intervention strategies (pp. 135-164). Emerald Group Publishing Limited.
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034